CLINICAL TRIAL: NCT03175744
Title: Prospective, Randomized, Multi-Center Study to Evaluate Treatment of Subjects With Occlusive Disease With a Novel Paclitaxel-Coated Angioplasty Balloon in Below-The-Knee (BTK) Arteries
Brief Title: Stellarex DCB Versus Standard Balloon Angioplasty for Treatment of Below-The-Knee (BTK) Arteries
Acronym: ILLUMENATE-BTK
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient enrollment impacted by COVID-19 pandemic and other business challenges. Patient enrollment discontinued, but follow-ups will continue according to protocol.
Sponsor: Spectranetics Corporation (Industry)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D032150
Record Dates: First submitted 2017-03-10; First posted 2017-06-05 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Stellarex DCB (Experimental): Spectranetics Stellarex Drug Coated Balloon
  Interventions: Device: Stellarex DCB
- PTA Catheter (Active Comparator): Standard Uncoated Balloon Angioplasty Catheter
  Interventions: Device: PTA Catheter

INTERVENTIONS:
Device: Stellarex DCB — Intervention with the Stellarex DCB
  Arms: Stellarex DCB
Device: PTA Catheter — Intervention with an uncoated Standard PTA
  Arms: PTA Catheter

SUMMARY:
The purpose is to demonstrate the safety and effectiveness of the Stellarex DCB for the treatment of stenosis or occlusions of below-the-knee arteries.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford Clinical Category 4-5
* Life expectancy > 1 year
* Significant stenosis ≥70%
* Patent inflow artery
* Target vessel(s) diameter between 2 and 4 mm
* Target vessel(s) reconstitute(s) at the ankle

Exclusion Criteria:

* Pregnant or planning to become pregnant
* History of stroke within 3 months
* Planned major amputation
* eGFR <30
* Acute limb ischemia
* Prior stent placement in target lesion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from Major Adverse Limb Event (MALE) | 30 days
  Composite of major amputation or major reintervention on a per patient basis
Freedom from Perioperative Death (POD) | 30 days
  Death on a per patient basis
Patency | 6 months
  Freedom from target lesion occlusion and clinically driven target lesion reintervention and freedom from major amputation on a per patient basis
Limb Salvage | 6 months
  Freedom from target lesion occlusion and clinically driven target lesion reintervention and freedom from major amputation on a per patient basis

SECONDARY OUTCOMES:
Clinically-driven target lesion revascularization | 6 months
  Rate of clinically-driven target lesion revascularization
Major adverse event rates | 6 months
  Composite rate of all-cause death, major amputation and clinically driven target lesion reintervention
Patency rate | 6 months
  Absence of target lesion occlusion and freedom from clinically-driven target lesion reintervention

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, MD, Principal Investigator — Lankenau Heart Institute; Mahmood K Razavi, MD, Principal Investigator — Vascular and Interventional Specialists of Orange; Dierk Scheinert, MD, Principal Investigator — University of Leipzig
Locations (21):
- United States (9):
  - St. Joseph Hospital, Orange, California
  - Bradenton Cardiology Center, Bradenton, Florida
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
- Australia (2):
  - Flinders Medical Center, Bedford Park
  - Sir Charles Gairdner Hospital, Perth
- Austria (2):
  - LKH Universitatsklinik Graz, Graz
  - Medizinische Universitat Wien, Vienna
- Belgium (3):
  - Imelda Ziekenhuis, Bonheiden
  - ZOL St. jan, Genk
  - University Hospital Gent, Ghent
- Germany (5):
  - Klinikum Hoschsauerland GmbH, Arnsberg
  - Universitats-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - SRH Klinikum Karlsbad, Karlsbad
  - Universitatsklink Leipzig, Leipzig
  - University Hospital of Tuebingen, Tübingen

IPD SHARING:
Plan to Share IPD: No